CLINICAL TRIAL: NCT04983264
Title: An Intrapatient Single Dose and Multiple Ascending Dose Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Pharmacodynamics of GBT021601, a Hemoglobin S Polymerization Inhibitor, in Participants With Sickle Cell Disease (SCD)
Brief Title: A Study to Evaluate GBT021601-012 Single Dose and Multiple Dose in Participants With Sickle Cell Disease (SCD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT021601-012; C5351002 (Other: Alias Study Number)
Record Dates: First submitted 2021-05-27; First posted 2021-07-30 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-dose Period (Part A) (Experimental): Refer to Study Description
  Interventions: Drug: GBT021601
- Multiple Ascending-dose Period (Part B and Part C) (Experimental): Refer to Study Description
  Interventions: Drug: GBT021601

INTERVENTIONS:
Drug: GBT021601 — Tablets and capsules which contain GBT021601 drug substance

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK), and pharmacodynamics (i.e., how the body absorbs, distributes, breaks down, and excretes) of GBT021601, a hemoglobin S (HbS) polymerization inhibitor, in participants with SCD, following single and multiple ascending doses.

DETAILED DESCRIPTION:
This is an open-label intrapatient single dose followed by a multiple dose escalation study in at least six (6) participants with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female with SCD
* Participants with SCD ages 18 to 60 years, inclusive.
* Participant has provided documented informed consent.
* Patients with stable and close to baseline hemoglobin value
* Patients on HU should be on stable dose for at least 90 days prior to signing ICF

Exclusion Criteria:

* Patients had more than 10 VOC within 12 months of screening
* Patients who are pregnant or nursing
* Patients who receive RBC transfusion therapy regularly or received an RBC transfusion for any reason within 60 days of signing the ICF
* Hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days of signing the ICF or within 24 days prior to Day 1 treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Advanced Pharma CR, LLC, Miami, Florida
  - Visionaries Clinical Research LLC, Atlanta, Georgia
  - Children's Healthcare of Atlanta AFLAC Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-012

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Single Dose Period: Participants received a single oral dose of GBT021601 100 mg on Day 1.
- Part B: Multiple Ascending- Dose Period: Participants received a loading dose on Day 56 (Week 8) followed by maintenance dose once weekly for up to 8 weeks. Dose administered in Part B of this study was in between a range of 50 mg to a maximum dose of 500 mg, based on the targeted % Hb occupancy of participants.
- Part C: Extended Treatment Period: Participants received a loading dose of 300 mg twice daily for 4 days followed by a maintenance dose of 150 mg once daily for up to 6 weeks.
Period: Part A: Single Dose Period
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Started (6) | 6 | 0 | 0
Completed (6) | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Multiple Dose Period
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Started | 0 | 6 | 0
Completed | 0 | 5 | 0
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Part C: Extended Treatment Period
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Started | 0 | 0 | 4 (Eligible participants from Part B entered to the extended treatment period.)
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Groups:
- Overall Study: All participants who received GBT021601 as single dose, multiple dose or extended treatment in Part A, Part B and Part C, respectively were included.
Arm/Group | Overall Study
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.2 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A treatment-emergent AE (TEAE) was an AE that occurs or worsens during the on-treatment period defined as the time from the first dose of study drug through minimum of 56 days after last dose of study treatment. A Serious Adverse Event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening experience (immediate risk of death); required inpatient hospitalization or prolongation if existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; was considered an important medical event. TEAEs and SAEs were reported for both Sickle Cell Disease (SCD) and non-SCD related events, in this outcome measure.
Time Frame: From first dose of study drug (Day 1) to at least 56 days after last dose of study drug (up to a maximum of 316 days)
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Participants
  TEAEs: SCD Related | 1 | 3 | 1
  SAEs: SCD Related | 0 | 2 | 0
  TEAEs: Non-SCD Related | 5 | 5 | 3
  SAEs: Non-SCD Related | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included were general appearance, head, ears, eyes, nose, throat, neck, skin, cardiovascular system, respiratory system, gastrointestinal system, musculoskeletal system, lymph nodes, and nervous system. Clinically significant physical examination abnormalities were considered as adverse events based on investigator's discretion.
Time Frame: Baseline (Day 1) up to at least 56 days after last dose of study drug (up to a maximum of 316 days)
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Multiple Ascending- Dose Period: Participants received a loading dose on Day 56 (Week 8) followed by maintenance dose once weekly for up to 8 weeks. Dose administered in Part B of this study was in between a range of 50 mg to a maximum dose of 500 mg, based on the % Hb occupancy of participants.
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Laboratory parameters included hematology(hemoglobin,hematocrit,red blood cell count,platelet count,white blood cell count,total neutrophils,eosinophils,monocytes,basophils,lymphocytes);blood chemistry(blood urea,nitrogen, creatinine,glucose,calcium,sodium,potassium,chloride,total bicarbonate,aspartate aminotransferase,alanine aminotransferase,total bilirubin,alkaline phosphatase,uric acid albumin,total protein);urinalysis(decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood,ketones, microscopy[urine tested positive for blood or protein]),urine drug screening:cannabinoids,amphetamines,methamphetamines,opiates,methadone,cocaine,benzodiazepines,phencyclidine,barbiturates,alcohol breath test. Hemoximetry RBC deformability,dense cells test; erythropoietin,follicle stimulating hormone,pregnancy test,Serology panel for HIV 1/2 antibody,Hepatitis A, B and C,SARS CoV-2.Clinical significance of any parameter was determined at the investigator's discretion.
Time Frame: Baseline (Day 1) up to at least 56 days after last dose of study drug (up to a maximum of 316 days)
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Participants | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs assessments included were systolic and diastolic blood pressure, heart rate, respiratory rate and body temperature. These measurements were taken after the participants had rested for at least 5 minutes in the supine position. Any clinically significant abnormal vital sign assessment required at least one repeat measurement. Clinical significance of any parameter was determined based on investigator's discretion.
Time Frame: Baseline (Day 1) up to at least 56 days after last dose of study drug (up to a maximum of 316 days)
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG)
Description: ECG values included here were Heart rate (HR), PR, QRS, QT, and QTcF intervals, interpretation of the tracings (eg, rhythm, presence of arrhythmia or conduction defects, any evidence of myocardial ischemia/infarction, or ST segment, T-wave, and U-wave abnormalities). Abnormal and clinically significant 12-lead ECG included QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 millisecond (ms), QRS interval >= 120 ms, PR interval > 220 ms, based on the average of triplicated ECG, assessed at Screening and Day-1. If any of these test results were out of range, then the test could be repeated once (in triplicate).
Time Frame: Baseline (Day 1) up to at least 56 days after last dose of study drug (up to a maximum of 316 days)
Population: Safety population was defined as all participants who received any amount of study drug (GBT021601).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Participants | 1 | 0 | 0

6. Secondary Outcome: Maximum GBT021601 Concentration (Cmax) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: Cmax was defined as the peak concentration observed directly from the experimental data without any interpolation.
Time Frame: Pre-dose, 0.25 hour (hr), 0.5 hr, 1 hr, 2 hrs, 4 hrs, 6 hrs, 8 hrs,12 hrs, 24 hrs, 36 hrs, 48 hrs, 72 hrs, 168 hrs, 336 hrs, 504 hrs, 672 hrs, 1008 hrs post-dose on Day 1
Population: Pharmacokinetic population was defined as all participants who received at least 1 dose of study drug (GBT021601) and had at least 1 plasma or whole blood concentration data point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
Microgram per milliliter (mcg/mL)
  Plasma | 1.01 (20.81)
  Whole Blood | 16.2 (25.90)
  RBC concentration | 69.2 (28.63)

7. Secondary Outcome: Maximum GBT021601 Concentration (Cmax) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part B
Description: Cmax was defined as the peak concentration observed directly from the experimental data without any interpolation.
Time Frame: Pre-dose, 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 56, 63, 70, 77, 84, 91, 98, 105, 112
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part B: Multiple Ascending- Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Plasma- Day 56 | 2.46 (15.27)
  Plasma- Day 63 | 1.28 (18.54)
  Plasma- Day 70 | 1.54 (32.36)
  Plasma- Day 77 | 1.17 (22.44)
  Plasma- Day 84 | 1.17 (19.75)
  Plasma- Day 91 | 5.15 (19.32)
  Plasma- Day 98 | 2.77 (16.41)
  Plasma- Day 105 | 2.96 (19.79)
  Plasma- Day 112 | 3.22 (15.50)
  Whole Blood- Day 56 | 40.9 (25.31)
  Whole Blood- Day 63 | 85.5 (40.91)
  Whole Blood- Day 70 | 80.3 (37.07)
  Whole Blood- Day 77 | 87.1 (41.84)
  Whole Blood- Day 84 | 89.1 (52.79)
  Whole Blood- Day 91 | 136 (41.37)
  Whole Blood- Day 98 | 201 (33.19)
  Whole Blood- Day 105 | 194 (44.14)
  Whole Blood- Day 112 | 200 (31.58)
  RBC concentration- Day 56 | 169 (25.28)
  RBC concentration- Day 63 | 366 (38.19)
  RBC concentration- Day 70 | 309 (38.95)
  RBC concentration- Day 77 | 337 (43.45)
  RBC concentration- Day 84 | 345 (50.80)
  RBC concentration- Day 91 | 522 (35.93)
  RBC concentration- Day 98 | 788 (25.66)
  RBC concentration- Day 105 | 748 (27.21)
  RBC concentration- Day 112 | 670 (33.48)

8. Secondary Outcome: Maximum GBT021601 Concentration (Cmax) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part C
Description: Cmax was defined as the peak concentration observed directly from the experimental data without any interpolation.
Time Frame: Pre-dose on Day 1, 14, 28, 42 and 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 28 and 42
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part C: Extended Treatment Period
Number analyzed (Participants) | 4
mcg/mL
  Plasma - Day 28 | 2.66 (78.79)
  Plasma - Day 42 | 4.25 (81.86)
  Whole Blood - Day 28 | 166 (126.31)
  Whole Blood - Day 42 | 175 (141.04)
  RBC concentration - Day 28 | 531 (105.76)
  RBC concentration - Day 42 | 540 (125.43)

9. Secondary Outcome: Minimum GBT021601 Concentration (Cmin) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part B
Description: Cmin was defined as the lowest concentration observed directly from the experimental data without any interpolation.
Time Frame: Pre-dose, 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 56, 63, 70, 77, 84, 91, 98, 105, 112
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part B: Multiple Ascending- Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Plasma- Day 63 | 0.97 (27.41)
  Plasma- Day 70 | 0.98 (22.18)
  Plasma- Day 77 | 0.90 (20.38)
  Plasma- Day 84 | 0.884 (21.58)
  Plasma- Day 91 | 0.90 (30.51)
  Plasma- Day 98 | 1.94 (24.77)
  Plasma- Day 105 | 1.84 (27.55)
  Plasma- Day 112 | 2.03 (24.43)
  Whole Blood- Day 63 | 62.6 (42.01)
  Whole Blood- Day 70 | 72.8 (36.26)
  Whole Blood- Day 77 | 77.4 (45.27)
  Whole Blood- Day 84 | 70.8 (67.54)
  Whole Blood- Day 91 | 76.5 (49.02)
  Whole Blood- Day 98 | 172 (43.11)
  Whole Blood- Day 105 | 161 (45.00)
  Whole Blood- Day 112 | 182 (31.55)
  RBC concentration- Day 63 | 267 (41.68)
  RBC concentration- Day 70 | 280 (38.56)
  RBC concentration- Day 77 | 299 (46.55)
  RBC concentration- Day 84 | 274 (65.32)
  RBC concentration- Day 91 | 299 (43.50)
  RBC concentration- Day 98 | 674 (34.28)
  RBC concentration- Day 105 | 621 (26.23)
  RBC concentration- Day 112 | 620 (34.72)

10. Secondary Outcome: Minimum GBT021601 Concentration (Cmin) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part C
Description: Cmin was defined as the lowest concentration observed directly from the experimental data without any interpolation.
Time Frame: Pre-dose on Day 1, 14, 28, 42 and 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 28 and 42
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part C: Extended Treatment Period
Number analyzed (Participants) | 4
mcg/mL
  Plasma - Day 28 | 1.54 (220.43)
  Plasma - Day 42 | 1.99 (264.95)
  Whole Blood - Day 28 | 122 (211.47)
  Whole Blood - Day 42 | 140 (217.11)
  RBC concentration - Day 28 | 392 (174.41)
  RBC concentration - Day 42 | 433 (187.77)

11. Secondary Outcome: Time to Attain Maximum Serum Concentration (Tmax) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: Maximum observed concentration was defined as the peak concentration observed directly from the experimental data without any interpolation. The time to the maximum observed concentration was defined as the time corresponding to Cmax.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
Hours
  Plasma | 1.50 [1.00 to 2.02]
  Whole Blood | 8.06 [6.00 to 35.92]
  RBC concentration | 8.06 [6.00 to 35.92]

12. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to the Next Dose (AUC0-tau) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: AUC0-tau was defined from time 0 to time of the last quantifiable concentration and was calculated using the linear or logarithmic trapezoid rule. AUCtau was calculated by using hours*microgram per milliliter (hr*mcg)/mL.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*mcg)/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
(hr*mcg)/mL
  Plasma | 67.102 (13.91)
  Whole Blood | 4597.8 (27.07)
  RBC concentration | 19627.6 (30.93)

13. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: AUCinf was defined as the area calculated by linear/log trapezoid rule from time 0 to infinity with the area extrapolated from the last quantifiable concentration to infinity.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*mcg)/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
(hr*mcg)/mL
  Plasma | 72.03 (16.43)
  Whole Blood | 4914.50 (29.55)
  RBC concentration | 234.08 (13.95)

14. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero up to Time 24 Hours (AUC 0-24) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: AUC0-24 was defined as the area under the free plasma concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Pre-dose, 0.25 hour (hr), 0.5 hr, 1 hr, 2 hrs, 4 hrs, 6 hrs, 8 hrs,12 hrs, 24 hrs post-dose on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*mcg)/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
(hr*mcg)/mL
  Plasma | 7.94 (12.11)
  Whole Blood | 322.0 (25.28)
  RBC concentration | 1363.3 (29.90)

15. Secondary Outcome: Apparent Oral Clearance (CL/F) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: CL/F was a quantitative measure of the rate at which a drug substance was removed from the blood. It was calculated as dose of GBT021601 by AUC from time 0 to infinity.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
Liter per hour
  Plasma | 1.39 (16.43)
  Whole Blood | 0.02 (29.55)
  RBC concentration | 0.004 (33.36)

16. Secondary Outcome: Terminal Elimination Half-Life (t1/2) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: t1/2 was the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
hr
  Plasma | 236.191 [187.44 to 313.49]
  Whole Blood | 230.908 [207.80 to 303.05]
  RBC concentration | 231.272 [206.58 to 302.82]

17. Secondary Outcome: Apparent Volume of Distribution (Vz/F) in Plasma, Whole Blood and Red Blood Cells (RBCs): Part A
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was determined based on the fraction absorbed.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
Liter
  Plasma | 480 (13.30)
  Whole Blood | 6.87 (22.56)
  RBC concentration | 1.61 (26.23)

18. Secondary Outcome: Percentage Hemoglobin Occupancy
Description: Percentage hemoglobin occupancy (%Hb Occupancy) refers to the proportion of hemoglobin molecules within red blood cells that were bound to study drug (GBT021601). Cmin and Cmax values was used to calculate %Hb occupancy: %Hb Occupancy = GBT021601*RBC per Mean Corpuscular Hemoglobin Concentration (MCHC).
Time Frame: Part A: Pre-dose,0.25,0.5,1,2,4, 6,8,12,24,36,48,72,168,336,504,672,1008 hrs on Day 1; Part B: Pre-dose,0.25 to 1,2 to 4 hrs post-dose on Day 56,63,70,77,84,91,98,105,112; Part C:Pre-dose on Day 1,14,28,42 and 0.25 to 1, 2 to 4 hrs post-dose on Day 28,42
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of Hemoglobin
Arm/Group | Part A: Single Dose Period | Part B: Multiple Ascending- Dose Period | Part C: Extended Treatment Period
Number analyzed (Participants) | 6 | 6 | 4
Percentage of Hemoglobin
  Part A: Cmax- Day 1: number analyzed (Participants) | 6 | 0 | 0
  Part A: Cmax- Day 1 | 3.36 (0.86) |  |
  Part B: Cmax- Day 56: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 56 |  | 8.15 (1.89) |
  Part B: Cmax - Day 63: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax - Day 63 |  | 18.15 (5.96) |
  Part B: Cmin- Day 63: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 63 |  | 13.40 (4.71) |
  Part B: Cmax- Day 70: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 70 |  | 15.50 (5.11) |
  Part B: Cmin- Day 70: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 70 |  | 14.03 (4.69) |
  Part B: Cmax- Day 77: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 77 |  | 17.03 (6.00) |
  Part B: Cmin- Day 77: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 77 |  | 15.25 (5.54) |
  Part B: Cmax- Day 84: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 84 |  | 17.66 (7.75) |
  Part B: Cmin- Day 84: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 84 |  | 14.57 (7.29) |
  Part B: Cmax- Day 91: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 91 |  | 25.71 (7.92) |
  Part B: Cmin- Day 91: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 91 |  | 15.02 (5.85) |
  Part B: Cmax- Day 98: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 98 |  | 38.00 (9.05) |
  Part B: Cmin- Day 98: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 98 |  | 33.04 (9.31) |
  Part B: Cmax- Day 105: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 105 |  | 36.11 (9.14) |
  Part B: Cmin- Day 105: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 105 |  | 29.89 (7.21) |
  Part B: Cmax- Day 112: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmax- Day 112 |  | 32.68 (9.33) |
  Part B: Cmin- Day 112: number analyzed (Participants) | 0 | 6 | 0
  Part B: Cmin- Day 112 |  | 30.32 (8.92) |
  Part C: Cmax- Day 28: number analyzed (Participants) | 0 | 0 | 4
  Part C: Cmax- Day 28 |  |  | 31.45 (17.97)
  Part C: Cmin- Day 28: number analyzed (Participants) | 0 | 0 | 4
  Part C: Cmin- Day 28 |  |  | 26.54 (16.96)
  Part C: Cmax- Day 42: number analyzed (Participants) | 0 | 0 | 4
  Part C: Cmax- Day 42 |  |  | 33.13 (19.12)
  Part C: Cmin- Day 42: number analyzed (Participants) | 0 | 0 | 4
  Part C: Cmin- Day 42 |  |  | 29.46 (18.09)

19. Secondary Outcome: Plasma Concentrations Versus Time Summary of GBT021601: Part A
Description: The plasma concentration versus time summary was measured by the amount of specific substance in the bloodstream over the specified timepoint.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Pre-dose | 0 (0)
  0.25 hour | 0.145 (0.137)
  0.5 hour | 0.617 (0.281)
  1 hour | 0.910 (0.312)
  2 hours | 0.821 (0.202)
  4 hours | 0.498 (0.150)
  6 hours | 0.350 (0.100)
  8 hours | 0.279 (0.737)
  12 hours | 0.228 (0.040)
  24 hours | 0.257 (0.120)
  36 hours | 0.333 (0.286)
  48 hours | 0.183 (0.067)
  72 hours | 0.138 (0.019)
  168 hours | 0.124 (0.020)
  336 hours | 0.0786 (0.016)
  504 hours | 0.047 (0.016)
  672 hours | 0.029 (0.137)
  1008 hours | 0.013 (0.007)

20. Secondary Outcome: Plasma Concentrations Versus Time Summary of GBT021601: Part B
Description: as for outcome 19
Time Frame: Pre-dose, 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 56, 63, 70, 77, 84, 91, 98, 105, 112, 140,168, 196, 218
Population: Pharmacokinetic population was defined as all participants who received at least 1 dose of study drug (GBT021601) and had at least 1 plasma or whole blood concentration data point. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: Multiple Ascending- Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Day 56: Pre-dose | 0.143 (0.351)
  Day 56 :0.25-1 hour | 1.163 (1.165)
  Day 56: 2-4 hours | 2.345 (0.3129)
  Day 63: Pre-dose | 1.015 (0.240)
  Day 63: 0.25-1 hour | 1.148 (0.268)
  Day 63: 2-4 hours | 1.250 (0.210)
  Day 70: Pre-dose | 1.003 (0.211)
  Day 70: 0.25-1 hour | 1.376 (0.653)
  Day 70: 2-4 hours | 1.415 (0.262)
  Day 77: Pre-dose | 0.937 (0.151)
  Day 77: 0.25-1 hour | 1.103 (0.318)
  Day 77: 2-4 hours | 1.173 (0.233)
  Day 84: Pre-dose | 0.918 (0.176)
  Day 84 :0.25-1 hour | 1.085 (0.284)
  Day 84: 2-4 hours | 1.097 (0.205)
  Day 91: Pre-dose | 0.941 (0.278)
  Day 91; 0.25-1 hour | 3.019 (2.225)
  Day 91: 2-4 hours | 4.990 (0.635)
  Day 98: Pre-dose | 2.118 (0.687)
  Day 98: 0.25-1 hour | 2.242 (0.398)
  Day 98: 2-4 hours | 2.580 (0.53933)
  Day 105: Pre-dose | 1.945 (0.570)
  Day 105: 0.25-1 hour | 2.147 (0.470)
  Day 105: 2-4 hours | 2.953 (0.642)
  Day 112 :Predose: number analyzed (Participants) | 4
  Day 112 :Predose | 2.095 (0.242)
  Day 112: 0.25-1 hour | 2.748 (0.824)
  Day 112: 2-4 hours | 2.905 (0.688)
  Day 140: 2-4 hours: number analyzed (Participants) | 5
  Day 140: 2-4 hours | 0.225 (0.0516)
  Day 168: 2-4 hours: number analyzed (Participants) | 4
  Day 168: 2-4 hours | 0.042 (0.026)
  Day 196: 2-4 hours: number analyzed (Participants) | 5
  Day 196: 2-4 hours | 0.005 (0.005)
  Day 218: 2-4 hours: number analyzed (Participants) | 5
  Day 218: 2-4 hours | 0.000 (0.001)

21. Secondary Outcome: Plasma Concentrations Versus Time Summary of GBT021601: Part C
Description: as for outcome 19
Time Frame: Pre-dose on Day 1, 14, 28, 42 and 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 28, 42, 70, 98
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part C: Extended Treatment Period
Number analyzed (Participants) | 4
mcg/mL
  Day 28: Pre-dose | 2.448 (1.786)
  Day 28: 4 hours | 2.991 (1.476)
  Day 42: Pre-dose | 3.621 (2.929)
  Day 42: 0.25-1 hour | 4.285 (2.785)
  Day 42: 2-4 hours | 4.485 (2.308)
  Day 70: 2-4 hours: number analyzed (Participants) | 3
  Day 70: 2-4 hours | 0.364 (0.101)
  Day 98: 2-4 hours: number analyzed (Participants) | 3
  Day 98: 2-4 hours | 0.034 (0.011)

22. Secondary Outcome: Whole Blood Concentrations Versus Time Summary of GBT021601: Part A
Description: The whole blood concentration versus time summary was measured to find concentration of various components in whole blood that changed over a specified period. This helped to monitor the dynamics of blood components such as hemoglobin levels, hematocrit, or glucose concentration over time.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Pre-dose | 0 (0)
  0.25 hour | 1.034 (0.876)
  0.5 hour | 4.775 (2.470)
  1 hour | 8.745 (3.833)
  2 hours | 12.710 (3.190)
  4 hours | 14.07 (2.917)
  6 hours | 14.44 (2.980)
  8 hours | 14.42 (2.861)
  12 hours | 14.45 (3.811)
  24 hours | 14.42 (3.220)
  36 hours | 15.41 (4.220)
  48 hours | 13.14 (2.895)
  72 hours | 12.42 (3.193)
  168 hours | 9.847 (2.562)
  336 hours | 5.282 (1.283)
  504 hours | 3.870 (1.071)
  672 hours | 2.138 (1.283)
  1008 hours | 0.943 (0.729)

23. Secondary Outcome: Whole Blood Concentrations Versus Time Summary of GBT021601: Part B
Description: as for outcome 22
Time Frame: Pre-dose, 0.25 hr to 1 hr, 2 to 4 hrs, post-dose on Day 56, 63, 70, 77, 84, 91, 98, 105, 112, 140,168, 196, 218
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: Multiple Ascending- Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Day 56: Pre-dose: number analyzed (Participants) | 5
  Day 56: Pre-dose | 0.071 (0.085)
  Day 56: 0.25-1 hour | 13.20 (13.601)
  Day 56: 2-4 hours | 41.23 (10.318)
  Day 63: Pre-dose | 74.32 (30.266)
  Day 63: 0.25-1 hour | 88.23 (33.335)
  Day 63: 2- 4 hours | 74.87 (19.748)
  Day 70: Pre-dose | 78.28 (24.403)
  Day 70: 0.25-1 hour | 81.00 (22.709)
  Day 70: 2-4 hours | 81.25 (25.669)
  Day 77: Pre-dose | 86.22 (30.703)
  Day 77: 0.25-1 hour | 87.33 (27.507)
  Day 77: 2- 4 hours | 88.68 (29.043)
  Day 84: Predose | 87.77 (43.076)
  Day 84 :0.25-1 hour | 88.97 (42.685)
  Day 84: 2-4 hours | 92.05 (36.530)
  Day 91: Pre-dose | 85.07 (32.859)
  Day 91; 0.25-1 hour | 102.4 (52.161)
  Day 91: 2-4 hours | 144.1 (47.113)
  Day 98: Pre-dose | 195.8 (61.979)
  Day 98: 0.25-1 hour | 188.8 (61.802)
  Day 98: 2-4 hours | 198.8 (49.301)
  Day 105: Pre-dose | 189.8 (56.672)
  Day 105: 0.25-1 hour | 178.9 (66.612)
  Day 105: 2-4 hours | 203.3 (74.923)
  Day 112: Pre-dose: number analyzed (Participants) | 4
  Day 112: Pre-dose | 195.0 (59.117)
  Day 112: 0.25-1 hour | 200.5 (57.263)
  Day 112: 2-4 hours | 198.5 (59.248)
  Day 140: 2-4 hours: number analyzed (Participants) | 5
  Day 140: 2-4 hours | 29.32 (20.149)
  Day 168: 2-4 hours: number analyzed (Participants) | 5
  Day 168: 2-4 hours | 3.082 (2.137)
  Day 196: 2-4 hours: number analyzed (Participants) | 5
  Day 196: 2-4 hours | 0.561 (0.560)
  Day 218: 2-4 hours: number analyzed (Participants) | 5
  Day 218: 2-4 hours | 0.108 (0.109)

24. Secondary Outcome: Whole Blood Concentrations Versus Time Summary of GBT021601: Part C
Description: as for outcome 22
Time Frame: Pre-dose on Day 1, 14, 28, 42 and 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 28, 42, 70, 98
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part C: Extended Treatment Period
Number analyzed (Participants) | 4
mcg/mL
  Day 28: Pre-dose | 202.2 (136.32)
  Day 28: 4 hours | 193.6 (106.16)
  Day 42: Pre-dose | 214.8 (131.21)
  Day 42: 0.25-1 hour | 213.5 (119.79)
  Day 42: 2- 4 hours | 229.9 (132.21)
  Day 70: 2-4 hours: number analyzed (Participants) | 3
  Day 70: 2-4 hours | 33.50 (2.553)
  Day 98: 2-4 hours: number analyzed (Participants) | 3
  Day 98: 2-4 hours | 3.310 (0.826)

25. Secondary Outcome: Red Blood Cell Concentrations Versus Time Summary of GBT021601: Part A
Description: The RBC concentration versus time summary was measured to identify quantity of RBC in a sample of blood over a specified duration. This analysis helped monitor RBC level over time.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: Single Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Pre-dose | 0 (0)
  0.25 hour | 3.989 (3.314)
  0.5 hour | 18.68 (10.413)
  1 hour | 34.84 (16.282)
  2 hours | 52.51 (14.931)
  4 hours | 59.50 (14.281)
  6 hours | 61.72 (15.356)
  8 hours | 61.68 (13.932)
  12 hours | 62.24 (18.340)
  24 hours | 61.92 (16.283)
  36 hours | 65.62 (18.780)
  48 hours | 56.60 (14.463)
  72 hours | 53.68 (15.728)
  168 hours | 42.41 (12.260)
  336 hours | 22.73 (6.316)
  504 hours | 16.65 (4.931)
  672 hours | 9.207 (5.652)
  1008 hours | 4.073 (3.186)

26. Secondary Outcome: Red Blood Cell Concentrations Versus Time Summary of GBT021601: Part B
Description: as for outcome 25
Time Frame: Pre-dose, 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 56, 63, 70, 77, 84, 91, 98, 105, 112, 140,168, 196, 218
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: Multiple Ascending- Dose Period
Number analyzed (Participants) | 6
mcg/mL
  Day 56: Pre-dose: number analyzed (Participants) | 5
  Day 56: Pre-dose | 0.120 (0.134)
  Day 56 :0.25-1 hour | 52.57 (53.388)
  Day 56: 2-4 hours | 170.8 (45.616)
  Day 63: Pre-dose | 317.4 (126.93)
  Day 63: 0.25-1 hour | 375.4 (134.89)
  Day 63: 2-4 hours | 318.6 (83.313)
  Day 70: Pre-dose | 304.7 (105.71)
  Day 70: 0.25-1 hour | 313.9 (97.320)
  Day 70: 2-4 hours | 314.7 (106.95)
  Day 77: Pre-dose | 335.9 (130.15)
  Day 77: 0.25-1 hour | 340.1 (118.67)
  Day 77: 2-4 hours | 343.8 (120.89)
  Day 84: Pre-dose | 338.6 (169.41)
  Day 84 :0.25-1 hour | 344.7 (170.26)
  Day 84: 2-4 hours | 356.0 (144.12)
  Day 91: Pre-dose | 329.0 (124.33)
  Day 91; 0.25-1 hour | 392.6 (197.92)
  Day 91: 2-4 hours | 547.7 (173.83)
  Day 98: Pre-dose | 753.5 (207.85)
  Day 98: 0.25-1 hour | 726.2 (215.42)
  Day 98: 2-4 hours | 768.9 (164.84)
  Day 105: Pre-dose | 711.7 (148.81)
  Day 105: 0.25-1 hour | 662.4 (190.38)
  Day 105: 2-4 hours | 752.8 (222.08)
  Day 112: Predose: number analyzed (Participants) | 4
  Day 112: Predose | 705.6 (209.26)
  Day 112: 0.25-1 hour | 674.3 (201.56)
  Day 112: 2-4 hours | 666.7 (206.56)
  Day 140: 2-4 hours: number analyzed (Participants) | 5
  Day 140: 2-4 hours | 120.8 (83.588)
  Day 168: 2-4 hours: number analyzed (Participants) | 5
  Day 168: 2-4 hours | 14.97 (9.339)
  Day 196: 2-4 hours: number analyzed (Participants) | 5
  Day 196: 2-4 hours | 2.326 (2.226)
  Day 218: 2-4 hours: number analyzed (Participants) | 5
  Day 218: 2-4 hours | 0.850 (0.539)

27. Secondary Outcome: Red Blood Cell Concentrations Versus Time Summary of GBT021601: Part C
Description: The RBC concentration versus time summary involved tracking a quantity of RBC in a sample of blood over a specified duration. This analysis helped to monitor RBC level over time.
Time Frame: Pre-dose on Day 1, 14, 28, 42 and 0.25 hr to 1 hr, 2 to 4 hrs post-dose on Day 28, 42, 70, 98
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part C: Extended Treatment Period
Number analyzed (Participants) | 4
mcg/mL
  Day 28: Pre-dose | 621.3 (428.95)
  Day 28: 4 hours | 594.4 (319.62)
  Day 42: Pre-dose | 642.4 (396.97)
  Day 42: 0.25-1 hour | 639.8 (361.11)
  Day 42: 2-4 hours | 691.1 (404.73)
  Day 70: 2-4 hours: number analyzed (Participants) | 3
  Day 70: 2-4 hours | 117.9 (20.028)
  Day 98: 2-4 hours: number analyzed (Participants) | 3
  Day 98: 2-4 hours | 12.74 (3.256)

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) up to at least 56 days after last dose of study drug (for a maximum of 316 days)
Description: Same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participants, or one participant may have experienced both serious and non-serious event during the study. AEs presented were related to both SCD and Non SCD related events.
Groups:
- Part A: Single Dose Period (SCD Related): Participants received a single oral dose of GBT021601 100 mg on Day 1 and had SCD related adverse events.
- Part B: Multiple Ascending- Dose Period (SCD Related): Participants received a loading dose on Day 56 (Week 8) followed by maintenance dose once weekly for up to 8 weeks. Dose administered in Part B of this study was in between a range of 50 mg to a maximum dose of 500 mg, based on the targeted % Hb occupancy of participants and had SCD related adverse events.
- Part C: Extended Treatment Period (SCD Related): Participants received a loading dose of 300 mg twice daily for 4 days followed by a maintenance dose of 150 mg once daily for up to 6 weeks and had SCD related adverse events.
- Part A: Single Dose Period (Non-SCD Related): Participants received a single oral dose of GBT021601 100 mg on Day 1 and had non-SCD related adverse events.
- Part B: Multiple Ascending- Dose Period (Non-SCD Related): Participants received a loading dose on Day 56 (Week 8) followed by maintenance dose once weekly for up to 8 weeks. Dose administered in Part B of this study was in between a range of 50 mg to a maximum dose of 500 mg, based on the targeted percentage Hemoglobin (% Hb) occupancy of participants and had non-SCD related adverse events.
- Part C: Extended Treatment Period (Non-SCD Related): Participants received a loading dose of 300 mg twice daily for 4 days followed by a maintenance dose of 150 mg once daily for up to 6 weeks and had non-SCD related adverse events.
Arm/Group | Part A: Single Dose Period (SCD Related) | Part B: Multiple Ascending- Dose Period (SCD Related) | Part C: Extended Treatment Period (SCD Related) | Part A: Single Dose Period (Non-SCD Related) | Part B: Multiple Ascending- Dose Period (Non-SCD Related) | Part C: Extended Treatment Period (Non-SCD Related)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/4 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/4 | 5/6 | 5/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Single Dose Period (SCD Related) (N=6) | Part B: Multiple Ascending- Dose Period (SCD Related) (N=6) | Part C: Extended Treatment Period (SCD Related) (N=4) | Part A: Single Dose Period (Non-SCD Related) (N=6) | Part B: Multiple Ascending- Dose Period (Non-SCD Related) (N=6) | Part C: Extended Treatment Period (Non-SCD Related) (N=4)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Single Dose Period (SCD Related) (N=6) | Part B: Multiple Ascending- Dose Period (SCD Related) (N=6) | Part C: Extended Treatment Period (SCD Related) (N=4) | Part A: Single Dose Period (Non-SCD Related) (N=6) | Part B: Multiple Ascending- Dose Period (Non-SCD Related) (N=6) | Part C: Extended Treatment Period (Non-SCD Related) (N=4)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT04983264/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT04983264/SAP_001.pdf